CLINICAL TRIAL: NCT01561716
Title: Is the Wii Fit / Wii Fit Plus Good Enough? A Comparison of the Energy Expenditure From Interactive Physical Activity Promoting Technology to Walking and Running
Brief Title: An Evaluation of the Energy Expenditure From Wii Fit Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ying Xian, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UL1RR024160/5-23087; UL1RR024160 (NIH)
Record Dates: First submitted 2012-03-14; First posted 2012-03-23 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Young Adults
Keywords: video games; energy expenditure; physical activity; exercise physiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Crossover sequence 1 (Experimental): Resting/Wii Fit Free Run/Wii Fit 3 bouts/treadmill
  Interventions: Device: Wii Fit
- Crossover sequence 2 (Experimental): Resting/Wii Fit Free Run/treadmill/Wii Fit 3 bouts
  Interventions: Device: Wii Fit
- Crossover sequence 3 (Experimental): Resting/Wii Fit 3 bouts/Wii Fit Free Run/treadmill
  Interventions: Device: Wii Fit
- Crossover sequence 4 (Experimental): Resting/Wii Fit 3 bouts/treadmill/Wii Fit Free Run
  Interventions: Device: Wii Fit
- Crossover sequence 5 (Experimental): Resting/treadmill/Wii Fit Free Run/Wii Fit 3 bouts
  Interventions: Device: Wii Fit
- Crossover sequence 6 (Experimental): Resting/treadmill/Wii Fit 3 bouts/Wii Fit Free Run
  Interventions: Device: Wii Fit

INTERVENTIONS:
Device: Wii Fit — This is a randomized, crossover study to evaluate the energy expenditure associated with Wii Fit games. After the baseline resting energy expenditure assessment, each participant complete the following physical activities on separate days in a random order, (1) 30-minute Wii Fit Aerobics Free Run, (2) 3 bouts of Wii Fit Aerobics (Advanced Step, Super Hula Hoop, and Rhythm Boxing in a random order) each lasting 10 minutes, and (3) 30-minute treadmill running/walking.

SUMMARY:
The purpose of this study is to provide energy expenditure data on Wii Fit / Wii Fit Plus games as compared with resting and treadmill walking/running.

DETAILED DESCRIPTION:
Increasing physical activity and, consequently, increasing energy expenditure and reducing obesity are among the highest public health priorities in the U.S. because physical inactivity negatively affects a wide variety of medical conditions (e.g., metabolic syndromes, cardiovascular disease). Research has shown that a major contributor to physical inactivity is the sedentary behavior induced by increased use of computer and video games. However, some of the newer generations of game consoles such as the Nintendo Wii market their product for its physical activity promoting features. Nintendo's recent release of Wii Fit / Wii Fit Plus uses a balance board and is the first game in which whole-body movements closely mirror that of the actual activity. As the use of these gaming systems may be more enjoyable modes of promoting physical activity than the traditional treadmill exercise, respondents may in turn exercise more regularly and for longer periods of time. To the best of the investigators' knowledge, no studies exist that demonstrate the energy expenditure of the Wii Fit / Wii Fit Plus among adults, or the Wii Fit / Wii Fit Plus compared to other forms of aerobic exercise such as walking and running. This study will provide preliminary data for future external grant applications comparing the energy expenditure of different physical activity conditions employing cutting-edge interactive physical activity promoting technology among adults. The potential contributions of the Wii Fit / Wii Fit Plus to promote healthy behaviors by being an alternative form of physical activity may be particularly informative for people who are unable to meet the national public health recommendations due to personal, health, safety or environmental concerns.

ELIGIBILITY:
Inclusion Criteria:

* No chronic disease by self-report (e.g. cardiovascular, renal, hepatic, neurodegenerative, neoplastic, metabolic {diabetes}, hypertension).
* Between the ages of 20-35.
* Normal BMI (BMI between 18.5 and 24.9).
* Not a current nicotine user.
* Demonstrates capacity for giving informed consent. Willing to participate by providing informed consent and committing to complete the study.

Exclusion Criteria:

* NA

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel D Fernandez, MD, PhD, MPH, Study Chair — University of Rochester; Ying Xian, MD, PhD, Principal Investigator — Duke Clinical Research Institute; Lisa Kakinami, PhD, Principal Investigator — McGill University
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty young healthy volunteers were enrolled in this randomized, crossover trial to examine the energy expenditure associated with Wii Fit and treadmill walking/running compared to sedentary resting between September 2009 and April 2010. Recruitment flyers were placed in the University of Rochester, Strong Memorial Hospital.
Pre-assignment Details: Each participant was assigned to a crossover sequence based on a computer generated randomization schedule using SAS 9.2. A washout period of at least 24 hours separated each study session.
Period: Overall Study
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 5 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (4.4) | 27.8 (4.0) | 26.4 (2.4) | 30.1 (2.4) | 28.9 (2.8) | 27.7 (3.7) | 28.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 2 | 2 | 5 | 21
  Male | 1 | 2 | 0 | 3 | 3 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure
Description: Energy expenditure is measured using continuous, computerized open-circuit indirect calorimetry (oxygen consumption and carbon dioxide production) and converted to metabolic equivalents (METs).
Time Frame: 30 min continuous monitoring at rest and during each physical activity
Measure: Mean (Standard Deviation); unit: METs
Groups:
- At Rest: Energy expenditure at rest
- Wii Fit Free Run: Energy expenditure during 30 min Wii Fit Free Run
- Wii Fit Super Hula Hoop: Energy expenditure during 10 min Wii Fit Super Hula Hoop
- Wii Fit Advanced Steps: Energy expenditure during 10 min Wii Fit Advanced Steps
- Wii Fit Rhythm Boxing: Energy expenditure during 10 min Wii Fit Rhythm Boxing
- Treadmill Running/Walking: Energy expenditure during 30 min treadmill running/walking
Arm/Group | At Rest | Wii Fit Free Run | Wii Fit Super Hula Hoop | Wii Fit Advanced Steps | Wii Fit Rhythm Boxing | Treadmill Running/Walking
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30
METs | 0.9 (0.1) | 5.0 (1.4) | 3.9 (1.3) | 3.8 (2.0) | 4.1 (0.9) | 8.0 (2.2)

ADVERSE EVENTS:
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The lab staffs that administrated the tests were not blinded to the order of the randomization, nor were they blinded to the results of the test. Thus, our study is subjected to observer and measurement biases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No